CLINICAL TRIAL: NCT01398098
Title: Gastric Emptying Time Assessment During Bowel Preparation With COLOKIT®
Brief Title: Measurement of Gastric Emptying During and After COLOKIT® Intake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Mayoly Spindler (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FCOL 111; 2011-002953-80 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-20 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Colonoscopy
MeSH Terms: interventions — sodium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COLOKIT® (Experimental)
  Interventions: Drug: Sodium phosphate

INTERVENTIONS:
Drug: Sodium phosphate — 32 tablets

SUMMARY:
Ultra-sound study to assess changes in intragastric volume after bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Subject who signed an informed consent to participate in the trial.
* Subject affiliated with Social Security
* Men and women aged 18 to 75 years.
* Subject with an indication of scheduled outpatient colonoscopy.
* colonoscopy performed within six hours after the second sequence COLOKIT®.
* Subject able to swallow tablets.

Exclusion Criteria:

1. Women pregnant or likely to be (without contraception) or nursing.
2. Subject having any of the following diseases or conditions:

   * allergy or hypersensitivity to the product tested or any of its excipients,
   * nausea, vomiting or abdominal pain,
   * clinically significant renal failure,
   * primary hyperparathyroidism associated with hypercalcemia,
   * congestive heart failure,
   * ascites,
   * a known or suspected bowel obstruction,
   * megacolon (congenital or acquired)
   * intestinal perforation,
   * ileus,
   * an inflammatory disease or suspected inflammatory bowel disease,
   * swallowing disorders,
   * known digestive motor disorders (gastroparesis, scleroderma, mega-esophagus),
   * diabetes mellitus (insulin or non insulin-dependent)
   * a history of gastric surgery (partial or total)
   * a contraindication to the anesthesia required for the completion of the colonoscopy,
   * Any clinical condition which, in the opinion of the investigator, would not allow the subject to perform the test in good conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a residual antral volume lower than 20 mL | after 2nd treatment regimen intake

SECONDARY OUTCOMES:
Adverse events | After drug intake
Acceptability of COLOKIT®. | After drug intake
Colonoscopy results | After colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas CHAUSSADE, Professor, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Derived] Coriat R, Polin V, Oudjit A, Henri F, Dhooge M, Leblanc S, Delchambre C, Esch A, Tabouret T, Barret M, Prat F, Chaussade S. Gastric emptying evaluation by ultrasound prior colonoscopy: an easy tool following bowel preparation. World J Gastroenterol. 2014 Oct 7;20(37):13591-8. doi: 10.3748/wjg.v20.i37.13591. PMID 25309090